CLINICAL TRIAL: NCT03797456
Title: A Multicenter, Open-label Study to Evaluate the Safety and Efficacy of ICP-022 in Patients With Relapsed/Refractory Marginal Zone Lymphoma (MZL)
Brief Title: A Study to Evaluate ICP-022 in Patients With R/R Marginal Zone Lymphoma (MZL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00104
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: MZL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-022 (Experimental)
  Interventions: Drug: ICP-022

INTERVENTIONS:
Drug: ICP-022 — ICP-022 (tablets, 50 mg) is given orally at the dose of 150 mg/day from day 1 to day 28 of each cycle for up to a total of 6 cycles or until progression.

SUMMARY:
The phase II clinical study is to investigate the safety, tolerability, efficacy and pharmacokinetics of ICP-022.

Safety, tolerability evaluation, and anti-tumor effects of ICP-022 in Chinese patients with R/R MZL will be evaluated in approximately 110 subjects. Pharmacokinetics of ICP-022 will be evaluated in approximately 20 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 75 years old
* Histologically confirmed marginal zone lymphoma (MZL), and at least one measurable tumor of greater than 1.5 centimeter outside of the spleen
* Subjects with refractory or relapsed MZL who has received at least 1 but no more than 4 prior therapies for MZL
* ECOG performance status of 0-2
* Documented failure to achieve at least partial response (PR) or documented disease progression after response to the most recent treatment regimen
* Subjects who have indications for treatment (threatened end-organ function, bulky disease >5cm, symptoms, steady progression, wish to treat)
* Subjects meet the following laboratory parameters:

  1. Absolute neutrophil count (ANC) ≥ 1.5×109/L Platelet count ≥ 75×109/L, independent of growth factor support within 7 days of the first dose with study drug, Hemoglobin ≥ 75 g/L; ANC ≥ 1.0×109/L, Platelet count ≥ 50×109/L, Hemoglobin ≥ 50 g/L; if bone marrow involvement
  2. Total bilirubin ≤ 1.5× ULN; AST or ALT ≤ 2× ULN; Creatinine ≤ 1.5× ULN; Amylase ≤ ULN and Lipase ≤ ULN
  3. International normalized ratio (INR) ≤ 1.5 ULN
* Life expectancy ≥ 3 months
* Able to provide signed written informed consent

Exclusion Criteria:

* History of other active malignancies within 5 years of study entry, unless cured without evidence of relapse or metastasis
* Current or history of lymphoma involved central nervous system
* Prior corticosteroids (at dosages equivalent to prednisone > 20 mg/day) given with anti-neoplastic intent within 7 days, prior chemotherapy, targeted therapy, radiation therapy, or antibody-based therapies or anti-cancer TCM within 4 weeks of the start of study drug
* Non-hematological toxicity must recover to ≤ Grade 1 from prior anti-cancer therapy (except for alopecia)
* Current clinically significant cardiovascular disease including:

  * Any class 3 or 4 cardiac disease such as arrhythmia, congestive heart failure or myocardial infarction defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction (LVEF) < 50%
  * Primary cardiomyopathy
  * Clinical significant QTc prolong history or QTc>470ms (female) QTc>450ms (male)
  * Uncontrolled hypertension
* Known active bleeding within 2 months of screening or currently taking anticoagulant/antiplatelet drugs
* Urine protein ≥ 2+ and quantitation ≥ 2g/24hours
* History of deep vein thrombosis or pulmonary embolism
* Toxicity must be recovered to ≤ Grade 1 from prior anti-cancer therapy
* Disease significantly affecting gastrointestinal function such as dysphagia, chronic diarrhea, intestinal obstruction, or resection of the stomach
* Prior organ or hematopoietic stem cell transplant
* Major surgery within 6 weeks of screening, except for diagnostic test or vascular access setup
* Known active infection with HBV, HCV or HIV or any uncontrolled active systemic infection
* Any history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe lung function impairment
* Prior exposure to a BTK or BCR pathway inhibitor (PI3K or Syk) and BCL-2 inhibitor
* Suitable and ready for allogeneic stem cell transplant
* Inability to comply with study procedures
* Drug abuser or alcoholics
* Lactating or pregnant women, or women who will not use contraception during the study and for 180 days after the last dose of study drug if sexually active and able to bear children
* Requires treatment with moderate or strong cytochrome P450 family 3, subfamily A (CYP3A) inhibitors or strong CYP3A inducers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 3 years
  The efficacy measured by overall response rate (ORR) in Part II according to the 2014 International Working Group NHL

SECONDARY OUTCOMES:
Occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria in Part I | Up to 3 years
  The safety of ICP-022 measured by the occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria in Part I
Progressioin free survival (PFS) | Up to 3 years
  Progression free survival (PFS) is defined as the time from registration to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
Duration of Response (DR) | Up to 3 years
  Duration of response as defined as the period from the first response (at least PR) to treatment until evidence of disease progression, relapse or death of any cause. Patients alive without progression and relapse will be censored at the latest tumor assessment date or the stopping date.
Overall survival (OS) | Up to 3 years
  Overall survival is defined as the period from the induction registration to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
Area under the concentration time curve up to the time "t" (AUC(0-t)) | up to 4 weeks
  Area under the concentration time curve up to the time "t" (AUC(0-t)) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.
Maximum plasma drug concentrations (Cmax) | up to 4 weeks
  Individual plasma concentrations of ICP-022 will be measured and Cmax will be calculated with noncompartmental analysis using WinNonlin.
Time of maximum plasma drug concentrations (Tmax) | up to 4 weeks
  Time of maximum plasma drug concentrations (Tmax) of ICP-022 will be recorded.
Apparent half-life for designated elimination phases (t½) | up to 4 weeks
  Apparent half-life for designated elimination phases (t½) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.
Area under the concentration time curve up to the last data point above LOQ (AUC(last)) | up to 4 weeks
  Area under the concentration time curve up to the last data point above LOQ (AUC(last)) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (32):
- China (32):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Anhui Cancer Hospital, Hefei, Anhui
  - Chinese People's Liberation Army General Hospital Fifth Medical Center, Beijing, Beijing Municipality
  - Peking university People's Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Union Hospital Affiliated to Fujian Medical University, Fuzhou, Fujian
  - The Second Hospital of Lanzhou University, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Shandong Provincial Hospital, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Cancer Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Hematology Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang University Medical School affiliated to the first Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No